CLINICAL TRIAL: NCT01476345
Title: Bioequivalence Study Comparing the Pharmacokinetics and Pharmacodynamics of LY2963016 With Insulin Glargine in Healthy Volunteers
Brief Title: A Study to Compare the Pharmacokinetics and Pharmacodynamics of LY2963016 to Lantus in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: 13711; I4L-MC-ABEA (Other: Eli Lilly and Company)
Record Dates: First submitted 2011-10-05; First posted 2011-11-22 (Estimated); Results first posted 2014-10-07 (Estimated); Last update posted 2014-10-07 (Estimated); Status verified 2014-10

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — LY2963016 insulin glargine; Insulin Glargine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- LY2963016 (Experimental): A single 0.5 units/kilogram (U/kg) dose of LY2963016 administered subcutaneously followed by minimum washout interval of 7 days.
  Interventions: Drug: LY2963016
- Lantus (Experimental): A single 0.5 U/kg dose of Lantus administered subcutaneously followed by minimum washout interval of 7 days.
  Interventions: Drug: Lantus

INTERVENTIONS:
Drug: LY2963016 — Administered subcutaneously
  Arms: LY2963016
Drug: Lantus — Administered subcutaneously
  Arms: Lantus

SUMMARY:
The purposes of this study are to determine the pharmacokinetics and pharmacodynamics of LY2963016 compared to those of basal insulin. The study will also gather information on the safety and tolerability of LY2963016 in healthy participants.

Each study period will be approximately 8.5 days (1.5 days for treatment and 7 day washout period). There are 4 study periods.

ELIGIBILITY:
Inclusion Criteria:

* are overtly healthy males or females, as determined by medical history and physical examination

  * male participants: agree to use a reliable method of birth control during the study.
  * female participants of child-bearing potential must test negative for pregnancy at the time of enrollment and agree to either abstain from sexual activity or to use a medically accepted means of contraception when engaging in sexual intercourse throughout the study, or female participants not of child-bearing potential due to surgical sterilization or menopause
* have a body weight of at least 55 kilograms (kg), and body mass index (BMI) of 18.5 to 32.0 kilograms/square meter (kg/m²)
* have clinical laboratory test results within normal reference range for the population
* have venous access sufficient to allow for blood sampling
* are reliable and willing to make themselves available for the duration of the study and are willing to follow study procedures
* have given written informed consent
* participants should have a normal oral glucose tolerance test

Exclusion Criteria:

* are currently enrolled in, have completed or discontinued within the last 30 days from, a clinical trial involving an investigational product other than the investigational product used in this study; or are concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study
* have known allergies to heparin, insulin glargine, related compounds or any components of the formulation
* are persons who have previously received the investigational product in this study, have completed or withdrawn from this study or any other study investigating LY2963016
* have an abnormality in the 12-lead electrocardiogram (ECG) that, in the opinion of the investigator, increases the risks associated with participating in the study
* have an abnormal blood pressure as determined by the investigator
* have a significant history or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, haematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the study medication
* show evidence of significant active neuropsychiatric disease
* regularly use known drugs of abuse and/or show positive findings on urinary drug screening
* show evidence of human immunodeficiency virus (HIV) infection and/or positive human HIV antibodies
* show evidence of hepatitis C and/or positive hepatitis C antibody
* show evidence of hepatitis B and/or positive hepatitis B surface antigen
* are women with a positive pregnancy test or women who are lactating
* intend to use over-the-counter or prescription medication
* have donated blood of more than 500 milliliters (mL) within the last 56 days before dosing of Period 1
* have an average weekly alcohol intake that exceeds 21 units per week (males) and 14 units per week (females), or are unwilling to stop alcohol consumption for 24 hours before dosing and throughout the duration of each study period
* smoke more than 10 cigarettes (or equivalent other tobacco products) per day
* have a fasting blood glucose > 5.5 millimoles/Liter (mmol/L) [>99 milligrams/deciliter (mg/dL)]at screening
* have a positive test for anti-LY2963016 or anti-glargine antibodies

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2011-11; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bloemfontein, South Africa

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was a randomized, 2-sequence, 4-period, crossover study.
Groups:
- LY/Lantus/LY/Lantus: Sequence 1: A single 0.5 units/kilogram (U/kg) dose of LY2963016 (LY) administered subcutaneously during Periods 1 and 3.
  A single 0.5 U/kg dose of Lantus administered subcutaneously during Periods 2 and 4.
  Minimum washout interval of 7 days between each period.
- Lantus/LY/Lantus/LY: Sequence 2: A single 0.5 U/kg dose of Lantus administered subcutaneously during Periods 1 and 3.
  A single 0.5 U/kg dose of LY2963016 administered subcutaneously during Periods 2 and 4.
  Minimum washout interval of 7 days between each period.
Period: Period 1
Arm/Group | LY/Lantus/LY/Lantus | Lantus/LY/Lantus/LY
Started | 40 | 40
Received at Least 1 Dose of Study Drug | 40 | 40
Completed | 40 | 40
Not Completed | 0 | 0
Period: Period 2
Arm/Group | LY/Lantus/LY/Lantus | Lantus/LY/Lantus/LY
Started | 40 | 40
Completed | 40 (1 did not enter Period 3 due to participant's decision.) | 40 (1 did not enter Period 3 due to participant's decision.)
Not Completed | 0 | 0
Period: Period 3
Arm/Group | LY/Lantus/LY/Lantus | Lantus/LY/Lantus/LY
Started | 39 | 39
Completed | 39 | 39
Not Completed | 0 | 0
Period: Period 4
Arm/Group | LY/Lantus/LY/Lantus | Lantus/LY/Lantus/LY
Started | 39 | 39
Completed | 39 | 39
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- All Participants: A single 0.5 units/kilogram (U/kg) dose of LY2963016 or a single 0.5 U/kg dose of Lantus administered subcutaneously followed by minimum washout interval of 7 days during 2 of 4 study periods in each sequence.
Arm/Group | All Participants
Number analyzed (Participants) | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.0 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 56
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 10
  White | 64
  More than one race | 6
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  South Africa | 80

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics: Area Under the Concentration-Time Curve From Time Zero to 24 Hours [AUC(0-24)] of LY2963016 and Lantus
Time Frame: 1 hour predose up to 24 hours postdose in all treatment periods
Population: All randomized participants who received at least 1 dose of study drug and had evaluable pharmacokinetic data to calculate AUC(0-24). Participants were analyzed based on the treatment they received.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picomoles*hour/Liter (pmol*h/L)
Groups:
- LY2963016: A single 0.5 units/kilogram (U/kg) dose of LY2963016 administered subcutaneously followed by minimum washout interval of 7 days during 2 of 4 study periods in each sequence.
- Lantus: A single 0.5 U/kg dose of Lantus administered subcutaneously followed by minimum washout interval of 7 days during 2 of 4 study periods in each sequence.
Arm/Group | LY2963016 | Lantus
Number analyzed (Participants) | 79 | 80
picomoles*hour/Liter (pmol*h/L) | 1810 (40) | 1980 (36)

2. Primary Outcome: Pharmacokinetics: Maximum Plasma Concentration (Cmax) of LY2963016 and Lantus
Time Frame: 1 hour predose up to 24 hours postdose in all treatment periods
Population: All randomized participants who received at least 1 dose of study drug and had evaluable pharmacokinetic data to calculate Cmax. Participants were analyzed based on the treatment they received.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picomoles/Liter (pmol/L)
Arm/Group | LY2963016 | Lantus
Number analyzed (Participants) | 80 | 80
picomoles/Liter (pmol/L) | 112 (39) | 119 (34)

3. Secondary Outcome: Maximum Glucose Infusion Rate (Rmax)
Description: Rmax is the maximum infusion rate of glucose administered intravenously needed to maintain target blood glucose level and is used to measure the study drug action over time as measured by the euglycaemic clamp procedure. During the euglycaemic clamp procedure, blood glucose concentrations are held constant after the administration of LY2963016 or Lantus by adjusting the exogenous glucose infusion rate. Data presented were adjusted by the body weight.
Time Frame: 1 hour predose up to 24 hours postdose in all treatment periods
Population: All randomized participants who received at least 1 dose of study drug and had evaluable data to calculate Rmax. Participants were analyzed based on the treatment they received.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milligrams/kilogram/minute (mg/kg/min)
Arm/Group | LY2963016 | Lantus
Number analyzed (Participants) | 80 | 80
milligrams/kilogram/minute (mg/kg/min) | 2.85 (46) | 2.88 (41)

4. Secondary Outcome: Total Amount of Glucose Infused (Gtot) Over the Duration of Clamp Procedure
Description: Gtot is the total glucose infusion over the clamp duration and is used to measure the study drug action over time as measured by the euglycaemic clamp procedure. During the euglycaemic clamp procedure, blood glucose concentrations are held constant after the administration of LY2963016 or Lantus by adjusting the exogenous glucose infusion rate. Data presented were adjusted by the body weight.
Time Frame: 1 hour predose up to 24 hours postdose in all treatment periods
Population: All randomized participants who received at least 1 dose of study drug and had evaluable data to calculate Gtot. Participants were analyzed based on the treatment they received.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milligrams/kilogram (mg/kg)
Arm/Group | LY2963016 | Lantus
Number analyzed (Participants) | 80 | 80
milligrams/kilogram (mg/kg) | 2580 (45) | 2710 (40)

ADVERSE EVENTS:
Arm/Group | LY2963016 | Lantus
Serious Adverse Events (participants affected / at risk) | 0/80 | 0/80
Other Adverse Events (participants affected / at risk) | 50/80 | 54/80
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | LY2963016 (N=80) | Lantus (N=80)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (5) | 5 (5)
Injection site erythema (General disorders) | 4 (4) | 2 (3)
Injection site pain (General disorders) | 5 (5) | 6 (7)
Procedural site reaction (Injury, poisoning and procedural complications) | 17 (21) | 17 (23)
Headache (Nervous system disorders) | 15 (19) | 25 (27)
Dysmenorrhoea (Reproductive system and breast disorders) | 1/24 (1) | 0/24 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators agreed to delay independently publishing or disclosing data, findings or conclusions from the study except as part of a multi-center publication. Upon study publication or if the draft publication is not produced within approximately 6 months of the final report of the study results, investigators may independently publish, subject to confidential information review/redaction by sponsor. The sponsor may request publication delay up to 90 days to seek patent protection.